CLINICAL TRIAL: NCT06484231
Title: Evaluation of the Effectiveness of Prophylactic Low Molecular Weight Heparin by Thromboelastography in Patients Who Underwent Lobectomy Due to Malignancy
Brief Title: Evaluation of the Effectiveness of Prophylactic LMWH by Thromboelastography
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gizem Kececi Ozgur, Principal investigator, Ege University
Other Study IDs: 22-AKD-64
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Malignancy
Keywords: malignancy; lobectomy; prophylaxis; thromboelastography
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to evaluate the necessity and effectiveness of using low molecular weight heparin (LMWH) for prophylaxis in the postoperative period in patients who underwent lobectomy due to malignancy, using thromboelastography.Blood samples taken from the patients before low molecular weight heparin prophylaxis (preoperative), before prophylaxis in the postoperative period (postoperative day 1) and after the start of postoperative prophylaxis (postoperative day 3) will be examined by thromboelastography.

DETAILED DESCRIPTION:
General characteristics of the patients such as age, gender, presence of comorbidities, smoking, type of operation and approach applied, operation duration, TEG measurements and postoperative complication development were recorded with case forms.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent lobectomy with thoracotomy or videothoracoscopy (VATS) due to malignancy (primary or secondary lung cancer)

Exclusion Criteria:

* Patients with a known diagnosis of bleeding or coagulation disorders
* Patients receiving anticoagulant and antiplatelet therapy in the preoperative period
* Patients who developed perioperative bleeding and therefore underwent perioperative blood and blood product replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent lobectomy due to malignancy
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
r time | 24 months
  'r time' value measured by thromboelastography
k time | 24 months
  'k time' value measured by thromboelastography
maximum amplitude (MA) | 24 months
  'MA' value measured by thromboelastography
angle a | 24 months
  'angle a' value measured by thromboelastography

SECONDARY OUTCOMES:
complications | 24 months
  development of complications

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Kececi Ozgur, Principal Investigator — Ege University Faculty of Medicine, Department of Thoracic Surgery
Locations (1):
- Ege University Faculty of Medicine, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moaad F, Zakhar B, Anton K, Moner M, Wisam S, Safy F, Igor W. Is LMWH Sufficient for Anticoagulant Prophylaxis in Bariatric Surgery? Prospective Study. Obes Surg. 2017 Sep;27(9):2331-2337. doi: 10.1007/s11695-017-2638-1. PMID 28326488
- [Background] Mukai M, Oka T. Mechanism and management of cancer-associated thrombosis. J Cardiol. 2018 Aug;72(2):89-93. doi: 10.1016/j.jjcc.2018.02.011. Epub 2018 Mar 24. PMID 29588087
- [Background] Wang Q, Ding J, Yang R. The venous thromboembolism prophylaxis in patients receiving thoracic surgery: A systematic review. Asia Pac J Clin Oncol. 2021 Oct;17(5):e142-e152. doi: 10.1111/ajco.13386. Epub 2020 Oct 2. PMID 33009716
- [Background] Klein SM, Slaughter TF, Vail PT, Ginsberg B, El-Moalem HE, Alexander R, D'Ercole F, Greengrass RA, Perumal TT, Welsby I, Gan TJ. Thromboelastography as a perioperative measure of anticoagulation resulting from low molecular weight heparin: a comparison with anti-Xa concentrations. Anesth Analg. 2000 Nov;91(5):1091-5. doi: 10.1097/00000539-200011000-00009. PMID 11049889
- [Background] Tekkesin N, Tekkesin M, Kaso G. Thromboelastography for the monitoring of the antithrombotic effect of low-molecular-weight heparin after major orthopedic surgery. Anatol J Cardiol. 2015 Nov;15(11):932-7. doi: 10.5152/akd.2014.5723. PMID 26574762
- [Background] Van PY, Cho SD, Underwood SJ, Morris MS, Watters JM, Schreiber MA. Thrombelastography versus AntiFactor Xa levels in the assessment of prophylactic-dose enoxaparin in critically ill patients. J Trauma. 2009 Jun;66(6):1509-15; discussion 1515-7. doi: 10.1097/TA.0b013e3181a51e33. PMID 19509608